CLINICAL TRIAL: NCT00001260
Title: Brain Procurement for the Human Brain Collection Core
Brief Title: Brain Tissue Collection for Neuropathological Studies
Status: Terminated | Type: Observational
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 900142; 90-M-0142
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Last update posted 2019-12-09 (Actual); Status verified 2017-06-16

CONDITIONS: Bipolar Disorder; Depression; Anxiety Disorders; Schizophrenia; Tourette's Syndrome; Brain Diseases
Keywords: Schizophrenia; Neuropathology; Neurochemistry; Substance Abuse; Bipolar Disorder; Aging; Normal Development; Depression; Anxiety Disorders; Suicide; Dementia; Neuropsychiatric Disorders; Tourette's Syndrome; Normal Controls
MeSH Terms: conditions — Bipolar Disorder; Depression; Anxiety Disorders; Schizophrenia; Tourette Syndrome; Brain Diseases; Substance-Related Disorders; Suicide; Dementia

SUMMARY:
The purpose of this study is to collect and study the brain tissue of deceased individuals to learn more about the nervous system and mental disorders. Information gained from donated tissue may lead to better treatments and potential cures for nervous system and mental disorders.

This study will ask relatives of deceased individuals to donate the brains of their deceased relatives to allow further study of neurological and psychiatric disorders. We do not accept prospective donations.

DETAILED DESCRIPTION:
The knowledge of how affected tissue deviates from normal control tissue is an integral part of fully understanding a neurological or psychiatric disorder. The purpose of this protocol is to establish a coordinating program with the Office of the Chief Medical Examiner in Washington, DC, the Virginia Office of the Chief Medical Examiner, Central District, and Virginia the Office of the Chief Medical Examiner, Northern District for the donation of brain tissue.

Dissected brain tissue from selected brain regions, including but not limited to the dorsolateral prefrontal cortex and hippocampal formation, will be assembled from large cohorts of normal controls and schizophrenic subjects. The expression of mRNA and protein for selected molecules, chosen on the basis of their genetic association with schizophrenia, will be measured with a variety of assays including but not limited to qPCR and Western blots.

Outcome measures are the statistical comparison within normal controls of mRNA and/or protein levels in groups segmented by genotype. Similar comparisons will be made between schizophrenic cohorts and normal controls, in a diagnosis by genotype analysis with an ANOVA, or when appropriate an ANCOVA (controlling for variables such as age, race, gender, and postmortem interval).

ELIGIBILITY:
* INCLUSION CRITERIA:

Brain tissue is needed from individuals suffering from a variety of neuropsychiatric disorders, especially schizophrenia, but also anxiety disorders, suicide, bipolar disorder, depression, Tourette's Syndrome, drug addictions (PCP, cocaine, alcohol, heroin or the like) and any form of dementia. In addition, brains from normal individuals without a history of neuropsychiatric disease will be needed for controls.

EXCLUSION CRITERIA:

No living subjects are enrolled in this protocol. Tissue is obtained after death, with the permission of next of kin, or from existing institutions with appropriate samples via an MTA or other applicable agreement.

Brain tissue is excluded from collection if there is a previously known history of strokes, lesions, or other major neuropathological abnormalities prior to the consenting process.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 2161 (Actual)
Dates: Start 1990-05-29; Study Completion 2017-06-16

CONTACTS AND LOCATIONS:
Overall Officials: Jose A Apud, M.D., Principal Investigator — National Institute of Mental Health (NIMH)
Locations (3):
- United States (3):
  - Office of the Chief Medical Examiner, Washington D.C., District of Columbia
  - National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland
  - Office of the Chief Medical Examiner, Fairfax, Virginia

REFERENCES:
- [Background] Meyer-Lindenberg A, Straub RE, Lipska BK, Verchinski BA, Goldberg T, Callicott JH, Egan MF, Huffaker SS, Mattay VS, Kolachana B, Kleinman JE, Weinberger DR. Genetic evidence implicating DARPP-32 in human frontostriatal structure, function, and cognition. J Clin Invest. 2007 Mar;117(3):672-82. doi: 10.1172/JCI30413. Epub 2007 Feb 8. PMID 17290303
- [Background] Law AJ, Lipska BK, Weickert CS, Hyde TM, Straub RE, Hashimoto R, Harrison PJ, Kleinman JE, Weinberger DR. Neuregulin 1 transcripts are differentially expressed in schizophrenia and regulated by 5' SNPs associated with the disease. Proc Natl Acad Sci U S A. 2006 Apr 25;103(17):6747-52. doi: 10.1073/pnas.0602002103. Epub 2006 Apr 17. PMID 16618933
- [Background] Egan MF, Straub RE, Goldberg TE, Yakub I, Callicott JH, Hariri AR, Mattay VS, Bertolino A, Hyde TM, Shannon-Weickert C, Akil M, Crook J, Vakkalanka RK, Balkissoon R, Gibbs RA, Kleinman JE, Weinberger DR. Variation in GRM3 affects cognition, prefrontal glutamate, and risk for schizophrenia. Proc Natl Acad Sci U S A. 2004 Aug 24;101(34):12604-9. doi: 10.1073/pnas.0405077101. Epub 2004 Aug 13. PMID 15310849
- [Derived] Bowen EFW, Burgess JL, Granger R, Kleinman JE, Rhodes CH. DLPFC transcriptome defines two molecular subtypes of schizophrenia. Transl Psychiatry. 2019 May 9;9(1):147. doi: 10.1038/s41398-019-0472-z. PMID 31073119
- [Derived] Mansur RB, Fries GR, Trevizol AP, Subramaniapillai M, Lovshin J, Lin K, Vinberg M, Ho RC, Brietzke E, McIntyre RS. The effect of body mass index on glucagon-like peptide receptor gene expression in the post mortem brain from individuals with mood and psychotic disorders. Eur Neuropsychopharmacol. 2019 Jan;29(1):137-146. doi: 10.1016/j.euroneuro.2018.10.007. Epub 2018 Nov 6. PMID 30409537
- [Derived] Mansur RB, Fries GR, Subramaniapillai M, Frangou S, De Felice FG, Rasgon N, McEwen B, Brietzke E, McIntyre RS. Expression of dopamine signaling genes in the post-mortem brain of individuals with mental illnesses is moderated by body mass index and mediated by insulin signaling genes. J Psychiatr Res. 2018 Dec;107:128-135. doi: 10.1016/j.jpsychires.2018.10.020. Epub 2018 Oct 27. PMID 30391805
- [Derived] Xiao X, Zhang C, Grigoroiu-Serbanescu M, Wang L, Li L, Zhou D, Yuan TF, Wang C, Chang H, Wu Y, Li Y, Wu DD, Yao YG, Li M. The cAMP responsive element-binding (CREB)-1 gene increases risk of major psychiatric disorders. Mol Psychiatry. 2018 Sep;23(9):1957-1967. doi: 10.1038/mp.2017.243. Epub 2017 Nov 21. PMID 29158582